CLINICAL TRIAL: NCT01761682
Title: Prospective Observational Cohort Registry for Patients With Acute Lymphoblastic Leukemia at Asan Medical Center
Brief Title: Acute Lymphoblastic Leukemia Registry at Asan Medical Center
Status: Terminated | Type: Observational
Why Stopped: The PI resigned the institute, and the rest investigators at the institute decided to terminate the study.
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Dae-Young Kim, Assistant Professor, Asan Medical Center
Other Study IDs: AMC-HEMREG-ALL
Record Dates: First submitted 2013-01-03; First posted 2013-01-07 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Leukemia, Acute Lymphoblastic; Precursor B-Cell Lymphoblastic Leukemia; Leukemia, Biphenotypic, Acute; Leukemia, Lymphoblastic, Acute, Philadelphia-Positive; Lymphoblastic Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor B-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Biphenotypic, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Bone marrow aspirate or peripheral blood (for its mononuclear cells) will be collected, processed, and cryopreserved for future analysis of DNA or cell culture. Acquisition of biospecimens will be proceeded if patient agree with the informed consent for donation of biospecimen to 'Asan Medical Center Biomaterial Resource Banking Center'. This registry data will be used as a basic demographic and clinical information for the biospecimens.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Ph-ALL: Diagnosed as ALL with Philadelphia-negative
  Interventions: Other: Diagnosed as ALL
- Ph+ALL: Diagnosed as ALL with Philadelphia-positive (including biphenotypic acute leukemia with Philadelphia-positive)
  Interventions: Other: Diagnosed as ALL
- Other ALL: Diagnosed as ALL of other type, including Burkitt leukemia
  Interventions: Other: Diagnosed as ALL

INTERVENTIONS:
Other: Diagnosed as ALL — All patients who will be enrolled in this prospective registry are confined to those who are diagnosed as acute lymphoblastic leukemia at Asan Medical Center, Seoul, Korea, from Jan 2013 till Dec 2047
  Other Names: Diagnosed as acute lymphoblastic leukemia

SUMMARY:
The investigators would like to propose a prospective longitudinal observational cohort study for patients who will be diagnosed and/or treated for acute lymphoblastic leukemia at Asan Medical Center, Seoul, Korea, to use the acquired data for fundamentals of other retrospective analysis.

DETAILED DESCRIPTION:
1. Acquisition of informed concent form
2. Data acquisition from medical record including

   * demographic / disease-associated factors
   * details of treatment, and its results
   * complications during treatment
   * genetic data
   * survival outcome (upto 10 years)
3. Accumulation of data for 30 years
4. Use of data for other retrospective analysis (including Asan Medical center Cell Banking basic data)

ELIGIBILITY:
Inclusion Criteria:

* All patients who are diagnosed and/or treated as acute lymphoblastic leukemia at Asan Medical Center (including biphenotypic acute leukemia with Philadelphila-positive, Burkitt leukemia/lymphoma)
* 15 years of age and over
* All patients who give written consent according to guidelines at Asan Medical Center committee on human research

Exclusion Criteria:

* Patients who refuse to give consent to registering

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are diagnosed and/or treated with acute lymphoblastic leukemia at Asan Medical Center, Seoul, Korea
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2013-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Overall survival | 10 year

SECONDARY OUTCOMES:
Event-free survival | 10 years
  Definition of events will be as 'relapse', 'death from any cause'. Relapse will be defined as hematologic relapse and molecular relapse, respectively when the patient is diagnosed as Philadelphia-positive acute lymphoblastic leukemia
Relapse-free survival | 10 years
  Relapse will be defined as hematologic relapse and molecular relapse, respectively when the patient is diagnosed as Philadelphia-positive acute lymphoblastic leukemia

CONTACTS AND LOCATIONS:
Overall Officials: Dae-Young Kim, MD, PhD, Principal Investigator — Associate Professor
Locations (1):
- Asan Medical Center, Seoul, South Korea